CLINICAL TRIAL: NCT03994380
Title: Use of DNAse in Neutrophilic Asthma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3030005151
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Neutrophilic Asthma
MeSH Terms: interventions — dornase alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): rhDNAse 2.5 mg nebulizer daily for 4 weeks
  Interventions: Drug: RhDNAse Inhalation Solution

INTERVENTIONS:
Drug: RhDNAse Inhalation Solution — rhDNAse 2.5 mg nebulizer daily for 4 weeks

SUMMARY:
In this pilot protocol, the researchers look to determine benefits from use of nebulized rh-DNase for 4 weeks in patients with neutrophilic asthma.

DETAILED DESCRIPTION:
Patients with asthma of a non-Th2 phenotype have few advanced therapeutic options if their asthma remains poorly controlled despite adherence to guideline-based therapy. Currently, no targeted biologic therapies are available for neutrophilic asthma. The role of Recombinant human deoxyriboneuclease (rhDNase) has not been investigated in refractory asthma. rhDNase cleaves extracellular DNA released by neutrophils and other granulocytes, thereby reducing the viscosity of mucus. It is known that patients with asthma have higher levels of extracellular DNA than normals; however, these levels are lower than DNA levels found in the sputum of patients with cystic fibrosis. The benefits of rhDNase in cystic fibrosis have been well described. In these patients, use of daily nebulized rhDNase has shown improvement in lung function and reduction in exacerbations. Very little is known about DNAse use in asthmatics. Case reports have shown benefit when used in acute asthma exacerbations, but there are no data on its use as a therapy for neutrophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

* i. Able to read and sign an Informed Consent Form (ICF)
* ii. At least Age 18
* iii. Diagnosis of Asthma with previous source documentation of PC 20 ≤ 16 mg/dl measured by FEV1 and/or reversibility with albuterol of ≥12% in FEV1
* iv. pre-bronchodilator Forced Vital Capacity (FVC) less than 85% predicted AND Serum total MMP9 ≥ 1800 (cut off determined by previous clinical investigation- Medimmune) OR serum IL-8> 20 pg/ml OR Sputum extracellular DNA ≥ 3.8 µg/mL OR Sputum Neutrophils > 40%

Exclusion Criteria:

* i. Pregnancy
* ii. Current smoker, smoking within the past year or pack/year history ≥ 10
* iii. Respiratory infection within past 6 weeks
* iv. Antibiotics within the past 4 weeks
* v. Active lung disease other than asthma
* vi. Cancer within the past 5 years (excluding basal cell skin cancer)
* vii. Chronic infection due to HIV, HBV, or HCV
* viii. Hematologic or autoimmune disease
* ix. Unable to safely undergo bronchoscopy as determined by primary or study doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Lung Function | 4 weeks
  FEV1
Symptom Control | 4 weeks
  Asthma Control Test

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States